CLINICAL TRIAL: NCT07369570
Title: A Prospective Study of the Evolution of Lesions in Repeated Biparametric Prostate Magnetic Resonance Imaging
Brief Title: Evolution of Lesions in Repeated Biparametric Prostate Magnetic Resonance Imaging
Acronym: REMRI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Juha Knaapila, MD, PhD, University of Eastern Finland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 218/13.00/2025
Record Dates: First submitted 2025-12-29; First posted 2026-01-27 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer (Diagnosis)
Keywords: prostate cancer; magnetic resonance imaging; mri; evolution; progression; pi-rads; significant; likert; pirads; biparametric; bpmri
MeSH Terms: conditions — Prostatic Neoplasms; Disease; Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Follow up arm (Experimental): Follow-up MRI and biopsy
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Biparametric follow-up prostate MRI and biopsies (systematic and targeted) for all study patients within one year, or earlier if the PSA value measured every three months increases by more than 50% from the baseline level in study inclusion, or if the physician has any other suspicion of high-risk prostate cancer.

SUMMARY:
The goal of this clinical trial is to prospectively investigate the evolution of lesions in biparametric magnetic resonance imaging (bpMRI) of the prostate in men with no clinically significant prostate cancer (csPCa) in their initial biopsy. The main questions it aims to answer are:

Does lesion progression in bpMRI predict a diagnosis of csPCa in per-protocol follow-up biopsies?

What are the radiological and clinical risk factors for csPCa in per-protocol follow-up biopsies?

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of a local prostate cancer
* Patient have 1-2 PI-RADS 3-5 lesion/lesions in biparametric prostate MRI, with no ISUP 2-5 prostate cancer in an initial systematic or lesion-targeted (at least two biopsy cores per lesion) biopsy
* Prostate biopsies can be taken via transrectal approach in an outpatient clinic
* An estimated life expentancy exceeding 10 years
* The patient is cooperative, fluent in Finnish and understands the significance of the study
* The patient signs an informed consent form approved by the ethics committee.

Exclusion Criteria:

* The patient had undergone prostate biopsies prior to the biopsies that led to recruitment for the current study.
* The physician's suspicion of a locally advanced or a high risk prostate cancer. Absolute exclusion criteria are PSA >20 ng/ml or T4 staged prostate finding MRI or clinical examination
* Seriuos infectious or non-infectious complication after initial biopsy
* Deep immunosuppression due to organ transplant, hematologic disease, or related causes.
* Any treatment given for prostate cancer diagnosed in initial biopsy
* Hip prosthesis or any other object in the pelvic area that affects high-quality MRI
* Claustrophobia or other absolute or relative contraindication for high-quality MRI

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-25 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
Evolution of MRI lesions | 3-12 months
  The evolution of biparametric prostate MRI findings during follow-up, assessed by the PRECISE score (1-5) using repeated biparametric prostate MRI-scan. Higher PRECISE score is associated with a higher risk of significant prostate cancer in prostate biopsy.
Evolution of MRI lesions | 3-12 months
  The evolution of biparametric prostate MRI findings (lesions) during follow-up, assessed by PI-RADS version 2.1 score (1-5), using repeated biparametric prostate MRI-scan. Higher PI-RADS score is associated with a higher risk of significant prostate cancer in prostate biopsy.
Evolution of MRI lesions | 3-12 months
  The evolution of biparametric prostate MRI findings during follow-up, assessed by lesional ADC value (s/mm2) using repeated biparametric prostate MRI-scan.
Evolution of MRI lesions | 3-12 months
  The evolution of biparametric prostate MRI lesions appearance in transrectal ultrasound (visible/non-visible) during follow up using repeated transrectal ultrasound.
Evolution of clinical factors | 3-12 months
  Assessment the effect of age (years) to the biopsy result in follow up prostate biopsy.
Evolution of clinical factors | 3-12 months
  Assessment the effect of PSA (ng/ml) level in baseline and during a follow up to the follow up prostate biopsy result using repeated laboratory tests and repeated prostate biopsy
Evolution of clinical factors | 3-12 months
  Assessment the effect of prostate size (g) to the biopsy result in follow up prostate biopsy. These factors will be measured by repeated biparametric prostate MRI scan and repeated prostate biopsy.
Evolution of clinical factors | 3-12 months
  Assessment the effect of PSA density (prostate size [g]/PSA value [ng/ml]) in baseline and follow up to the biopsy result in follow up prostate biopsy. These factors will be measured by repeated biparametric prostate MRI scan, repeated laboratory tests and repeated prostate biopsy.
Biopsy result during follow up | 3-12 months
  Amount of prostate cancer and prostate cancer upgrade/downgrade in repeated systematic and lesion targeted prostate biopsy during the follow up. Prostate biopsy result will be graded using ISUP Gleason Grade Group (benign, 1-5). Higher ISUP Gleason Grade Groups score is associated with a worse oncological outcomes.